CLINICAL TRIAL: NCT01758055
Title: Safety Study of Endobronchial Transplantation of Autologous Mesenchymal Stem Cells Derived Bone Marrow in Patients With Emphysema
Brief Title: Safety Study of Endobronchial Transplantation of Autologous Mesenchymal Stem Cells (MSCs) in Emphysema Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Arda Kiani (Other)
Collaborators: Royan Institute (Other Government)
Responsible Party: Sponsor-Investigator, Arda Kiani, Professor of Shahid Beheshti University, Masih Daneshvari Hospital
Organization: Masih Daneshvari Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: f-91-135
Record Dates: First submitted 2012-11-18; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-11

CONDITIONS: Emphysema
Keywords: Mesenchymal stem cell, emphysema, lung function
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous MSCs transplantation (Experimental): intra bronchial injection, Autologous MSCs transplantation derived bone marrow, 60millions cells, once
  Interventions: Biological: Autologous MSCs transplantation

INTERVENTIONS:
Biological: Autologous MSCs transplantation — Autologous mesenchymal stem cells derived bone marrow, bronchoscopy

SUMMARY:
The purpose of this study is evaluating the safety of endobronchial transplantation of autologous mesenchymal stem cells derived bone marrow in patients with emphysema.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a worldwide epidemic disease that the global prevalence of it was estimated to be approximately 210 million individuals and accounting for more than three million deaths annually. And currently, it is the fifth chief cause of death in the United State of America. COPD is characterized by chronic, irreversible inflammation of the airways and has two pathologic features, emphysema and bronchiolitis.

The most relevant feature in the lung emphysema is airflow limitation, resulting from the loss of alveolar wall and enlargement of alveolar space distal to the terminal bronchiole. Cigarette and air pollution are the most major factors for developing COPD. Unfortunately, aside from supplemental domiciliary oxygen for the small number of patients who demonstrate resting arterial hypoxemia and smoking cessation for continued smokers, there are no interventions that have been unequivocally shown to prolong survival in patients with COPD. In the preprocessing phase, patients will underwent a complete evaluation of the pulmonary function test with spirometer to measure the FEV1, FVC, FEV1/FVC, cardiac evaluation (clinical examination, six minute walk test, echocardiography TTE(transthoracic echocardiography ), and electrocardiography),chest X-ray, chest computed tomography scan (helical/high resolution),o2 saturation by oximeter, as well as routine laboratory tests (blood gas, urinalysis, coagulation, complete blood count (CBC), blood urea nitrogen, fasting glucose, creatinine, AST(aspartate aminotransferase), ALT(alanine aminotransferase), C-reactive protein, serology for hepatitis B and C, antihuman immunodeficiency virus, and treponemal test for syphilis (FTA-ABS)). The Dyspnea Scale Score test, modified according to the British MMRC, was also conducted, according to Mahler and Wells and Curley.And quality of life measures will assess according to SF-36(Medical Outcomes Study 36-Items Short-Form Health Survey) questioner.

Patients will taken to the operating room, placed in a prone position, and administer a spinal anesthesia. Approximately, 120 mL of bone marrow will aspirated from each puncture and after preparation about 60 million autologous MSCs will transplant by bronchoscopy into the endobronchial of these patients.

ELIGIBILITY:
Inclusion Criteria:

* • Inclusion criteria were as follows:

  * patients with moderate to severe emphysema that has a FEV1≤50% (approved by HRCT)
  * aged less than 70 years
  * no tobacco use for at least 12 months before the protocol application
  * no serious coronaropathy and/or ventricular dysfunction
  * no significant renal illness and/or hepatitis
  * EF(ejection fraction)>50%
  * Creatinine < 2
  * AST, ALT≤ 10 times of its normal basis

Exclusion Criteria:

* Exclusion criteria were as follows:

  * detected immunosuppressive illnesses
  * carrier of known neoplasias
  * pregnancy
  * limitation in daily physical activities
  * known case of diabetic disorders
  * modifying in his/her medical treatment regime in the past year

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
forced vital capacity( FVC), forced expiratory volume(FEV1), FEV1/FVC | Baseline and one year after procedure
  * A pulmonary function test that measures the volume and speed of inhaled air.
  * A pulmonary function test that measures the volume and speed of exhaled air.

SECONDARY OUTCOMES:
six minute walk test | Baseline and One year after procedure
  •A six minute walk test with treadmills

OTHER OUTCOMES:
oxygen saturation | Baseline and one year after procedure
  •An oximeter test for evaluating the oxygen saturation
Quality of life | Baseline and One year after procedure
  •A SF36 quality of life questioner for evaluating the quality of life
DLCO(diffusion capacity of lung for carbon monoxide) | Baseline and One year after procedure
  •Body Box device for evaluating diffusing capacity of the lung for carbon monoxide
CT scan | Baseline and One year after procedure
  •A CT scan for evaluating the changes
dyspnea score | Baseline and One year after procedure
  •A MMRC(modified medical research council) scale for evaluating the dyspnea score
Atrial blood gases test-PaO2(partial pressure of oxygen in blood) , PaCO2(partial pressure of carbon dioxide in blood) | Baseline and one year after procedure
  * presence of oxygen in blood gases
  * presence of carbon dioxide in blood gases
Infection | Baseline and one year after procedure
  •A CBC test for evaluating the infection

CONTACTS AND LOCATIONS:
Overall Officials: Arda Kiani, MD, pulmono, Study Director — Tracheal Diseases Research Center, Shahid Beheshti University of Medical Sciences, Tehran, Iran.; Naser Aghdami, MD,PHD, Study Director — Department of Regenerative Biomedicine and cell therapy,Cell science Research Center,Royan Institute for Stem Cell Biology and Technology,ACER,Tehran,Iran
Locations (1):
- Masih-Daneshvari Hospital, Tehran, Tehran Province, Iran